CLINICAL TRIAL: NCT01764035
Title: The Effects of Mindfulness on Disrupted Sleep in Bipolar Disorder
Brief Title: Mindfulness Therapy on Disrupted Sleep in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Thilo Deckersbach, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P002550
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Bipolar Disorder; Insomnia; Hypersomnia; Sleep Problems
Keywords: Psychotherapy; Bipolar Disorder; Sleep Problems; Insomnia; Hypersomnia; Mindfulness; Meditation; Sleep Disturbance
MeSH Terms: conditions — Bipolar Disorder; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Supportive Psychotherapy (SP) (Active Comparator): 30 people will be randomized to receive Brief Supportive Psychotherapy.
  Interventions: Behavioral: Brief Supportive Psychotherapy (SP)
- Body Scan (BS) Meditation Intervention (Experimental): 30 people will be randomized receive the Body Scan Meditation Intervention.
  Interventions: Behavioral: Body Scan (BS) Meditation Intervention

INTERVENTIONS:
Behavioral: Body Scan (BS) Meditation Intervention — This intervention consists of 4 individual 60-minute sessions (week 1, 2, 4, and 6) in which participants learn the body scan meditation exercise and practice it at home, daily, lying in bed at their usual bedtime after going to bed (and when waking up at night, unable to go back to sleep). The Body-Scan meditation consists of a 30-minute exercise during which participants are guided to focus their attention on certain parts of their body (e.g. toes, feet). The core skill involves gradually adopting an observant, non-judgmental, and accepting stance towards bodily sensations, including feelings and thoughts.
  Arms: Body Scan (BS) Meditation Intervention
Behavioral: Brief Supportive Psychotherapy (SP) — SP is a common form of non-specific psychotherapy available to patients with bipolar disorder in the community. It focuses on addressing a patient's current concerns, supporting a patient's adaptive coping skills, improving self-esteem, and expressing feelings and the therapeutic alliance. Using a conversational style, SP involves conveying empathy, validation, comforting and supporting patients in coping with distress about current life issues as well as providing encouragement and praise, clarification and opportunity to vent. SP will match BS in length, number of sessions and delivery schedule (four, 60-minute sessions, week 1, 2, 4, 6).
  Arms: Brief Supportive Psychotherapy (SP)

SUMMARY:
The investigators propose to investigate the efficacy of a brief (4-session) Body Scan (BS) meditation intervention for individuals with bipolar I disorder with insomnia (i.e. difficulties falling or staying asleep). The investigators will compare the Body Scan intervention with a 4-session brief supportive psychotherapy (SP) intervention. The investigators hypothesize that the Body Scan will improve objective sleep quantity and quality.

DETAILED DESCRIPTION:
This is the first evaluation of the efficacy of a mindfulness-based intervention for insomnia in bipolar disorder. It distills the findings from previous mindfulness-based interventions for other disorders that documented beneficial effects for sleep, by concentrating on the most active mindfulness ingredient for treating sleep (the Body Scan). To date, mindfulness based studies have focused on either subjective sleep reports or laboratory-based measures of sleep, both of which have long been called into question because of their lack of ecological validity. This study takes advantage of recent developments in ambulatory sleep monitoring by using the new, FDA approved M1 device, which assesses sleep objectively in a patient's home environment. The M1 device is also the only ambulatory sleep-monitoring device to date that simultaneously assesses both sleep quantity and quality. Finally, this study broadens the view above and beyond sleep and mood and investigates the impact on cognitive and sleep-related psychosocial functioning, both at the end of treatment as well as at a 3-month follow-up. Overall, this work could result in a brief, easy to administer, and easy to disseminate intervention for patients with bipolar disorder with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65
* DSM-IV diagnosis of bipolar I or II disorder
* HAM-D-17 score < 17 (i.e. low or no depressive symptoms)
* YMRS score < 8 (i.e. no or low manic symptoms)
* Optimized, stable maintenance pharmacotherapy at maximum tolerated dosages in accordance with the revised Texas Implementation of Medication Algorithm
* DSM-IV insomnia A and B criteria are met (i.e. difficulty initiating or maintaining sleep, for at least 1 month) as operationally defined by:

  1. Insomnia Severity Index score of > 15 (moderate clinical insomnia)
  2. M1 derived average actigraphic total sleep time < 6 hours, and < 40% average total sleep time in high frequency coupling, as measured with the M1 device over 5 days pre-randomization, corresponding to < 1SD below the mean of the M1 normative comparison sample of healthy control participants.

Exclusion Criteria:

* DSM-IV bipolar I disorder subtype rapid cycling
* DSM-IV manic or mixed episode in the past 2 months
* DSM-IV major depressive episode in the past 2 months
* Psychotropic medication not in accordance with the revised Texas Implementation of Medication Algorithm
* Pregnancy
* Medical illness or non-psychiatric medical treatment that is the likely cause of the sleep disturbance or interferes with study participation
* Neurologic disorder, previous ECT, or history of head trauma (i.e. known structural brain lesion)
* Current or past history of selected DSM-IV Axis I disorders other than bipolar disorder including: organic mental disorder, substance abuse within the past 12 months and/or history of substance abuse for > 1 year; past or current substance dependence (including alcohol), schizophrenia, delusional disorder, psychotic disorders not otherwise specified
* Axis I disorder that needs to be the primary focus of treatment (e.g. current DSM-IV anxiety disorder that disrupts sleep)
* Sleep apnea, restless leg syndrome, or narcolepsy
* Concurrent psychotherapy to BS or SP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | 8 weeks

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | 20 weeks
  Young Mania Rating Scale is an 11-item, clinician-rated measure that assesses the presence and severity of patient's current symptoms of mania.
Hamilton Depression Rating Inventory (HAM-D 17). | 20 weeks
  The HAM-D 17 is an established clinician-rated outcome measure in treatment trials for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Deckersbach, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States